CLINICAL TRIAL: NCT06000345
Title: Effect of Action Observation and Motor Imagery on Arthrogenic Muscle Inhibition of the Quadriceps in Patients With End-stage Knee Gonarthrosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLF22/07
Record Dates: First submitted 2023-08-03; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Knee Osteoarthritis; Arthrogenic Muscle Inhibitions
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AOT + MI group (Experimental): The AOT + MI group was shown a video (4 minutes) in which a subject (matched for age, sex, and limb affected) performed, in third person view, quadriceps concentric contractions for 2 minutes and isometric contractions for 2 minutes. The video contained visual elements indicating the maximality of the effort. After both concentric and isometric movement video the subjects performed a MI session (1 minute in length each), in which they were asked to imagine in first person the action previously observed in the video.
  Interventions: Other: AOT + MI
- Control group (Sham Comparator): The control group was shown a video of landscapes (4 minutes in length). Halfway through and at the end of the video they were asked to imagine what they had just seen for 1 minute.
  Interventions: Other: Control AOT + MI

INTERVENTIONS:
Other: AOT + MI — During the AOT session, the patients were shown a video containing motor contents. In particular, the video demonstrated quadriceps concentric and isometric contractions, presented in the third person perspective. At the conclusion of each video, the patients were asked to spend 1 minute imagining what they had just seen.
  Arms: AOT + MI group
Other: Control AOT + MI — The control group was shown a video of landscapes (4 minutes in length). Halfway through and at the end of the video they were asked to imagine what they had just seen for 1 minute.
  Arms: Control group

SUMMARY:
The study aims at evaluating the effects of one session of Action Observation Training (AOT) and Motor Imagery (MI) on arthrogenic muscle inhibition (AMI) of the quadriceps (QF) in subjects with end-stage gonarthrosis.

30 patients with end-stage knee osteoarthritis were enrolled. Patients were randomized in two groups (experimental group and control group).

Experimental group performed one 6-minutes AOT and MI session with motor content of concentric and isometric QF contractions, whereas control group underwent a 6-minute sham AOT and MI session. Every patient was evaluated to assess the percentage of AMI on the QF before (T0) and after (T1) the treatment following the gold standard Twitch Interpolated Technique.

DETAILED DESCRIPTION:
The study aims at evaluating the effects of one session of Action Observation Training (AOT) and Motor Imagery (MI) on arthrogenic muscle inhibition (AMI) of the quadriceps (QF) in subjects with end-stage gonarthrosis.

30 patients with end-stage knee osteoarthritis were enrolled. Patients were randomized in two groups (experimental group and control group).

Experimental group performed one AOT and MI session with motor content of concentric and isometric QF contractions, whereas control group underwent a 6-minute sham AOT and MI session. Every patient was evaluated to assess the percentage of AMI on the QF before (T0) and after (T1) the assigned treatment following the gold standard Twitch Interpolated Technique. Both groups sat on an isometric dynamometric chair (COR1, OT-Bioelettronica, Torino) with a load cell (FORZA, OT-Bioelettronica, Torino) designed to detect and map the strenght generated by the QF muscle. Upper body movements were limited by crossover shoulder harnesses, a belt across the abdomen and the subjects were asked to keep their arms crossed holding onto the harness while performing the evaluation.

Three large electrodes (10x13cm) were positioned over the quadriceps muscle belly. Two sEMG electrodes (FREEEMG, BTS, Italy) were positioned on the Vastus Medialis and Vastus Lateralis using the SENIAM protocol.

Right after the first evaluation (T0), both groups performed an AOT session. The experimental group was shown a video (4 minutes) in which a subject (matched for age, sex, and limb affected) performed, in third person view, quadriceps concentric contractions for 2 minutes and isometric contractions for 2 minutes. The video contained visual elements indicating the maximality of the effort. After both concentric movement video and isometric movement video the subjects performed a MI session (2 sessions, 1 minute in length each), in which they were asked to imagine in first person the action just seen in the video.

On the other hand, the control group was shown a video of landscapes (4 minutes in length). Halfway through and at the end of the video they were asked to imagine what they had just seen for 1 minute. After the session of AOT and MI (T1) both groups were re-evaluated in the same way as previously described.

ELIGIBILITY:
Inclusion Criteria:

* patients with end-stage knee ostheoarthritis undergoing primary total knee arthroplasty
* Active knee flexion > 45°

Exclusion Criteria:

* Previous lower limb orthopedic surgery
* Concomitant neurological, orthopedic, cardiovascular disorders
* Cognitive impairments or psychiatric disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-09-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes in arthrogenic muscle inhibition (estimated through Interpolated Twitch Technique) | 1- Before AOT+MI session; 2- Immediately after AOT+MI session
  Changes in arthrogenic muscle inhibition (AMI) of the quadriceps muscle before and after AOT and MI session on patients with advanced stage gonarthrosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Italy

IPD SHARING:
Plan to Share IPD: No